CLINICAL TRIAL: NCT05410223
Title: A Study on the Efficacy and Safety of Egg Yolk Antibody in Adjuvant Treatment of Helicobacter Pylori Infection
Brief Title: Efficacy and Safety Study of Egg Yolk Antibody in Adjuvant Treatment of Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xucanxia2020
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Egg yolk antibody; Helicobacter pylori rescue therapy; Helicobacter pylori therapy
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Furazolidone; Doxycycline; Bismuth

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- study group (Experimental): 14-days therapy of Yolk antibody and ilaprazole, clarithromycin/amoxicillin/furazolidone, doxycycline, bismuth
  Interventions: Drug: Yolk antibody and IIaprazole, Amoxicillin/ Clarithromycin/Furazolidone, Doxycycline, Bismuth
- control group (Active Comparator): 14-days therapy of ilaprazole, clarithromycin/amoxicillin/furazolidone, doxycycline, bismuth
  Interventions: Drug: IIaprazole, Amoxicillin/Clarithromycin/Furazolidone, Doxycycline, Bismuth
- the case group (Experimental): 14-days therapy of Yolk antibody and ilaprazole, clarithromycin/amoxicillin/furazolidone, doxycycline
  Interventions: Drug: Yolk antibody and IIaprazole, Amoxicillin/ Clarithromycin/Furazolidone, Doxycycline
- the control group (Active Comparator): 14-days therapy of ilaprazole, clarithromycin/amoxicillin/furazolidone, doxycycline, bismuth
  Interventions: Drug: IIaprazole, Amoxicillin/ Clarithromycin/Furazolidone, Doxycycline, Bismuth

INTERVENTIONS:
Drug: Yolk antibody and IIaprazole, Amoxicillin/ Clarithromycin/Furazolidone, Doxycycline, Bismuth — Yolk antibody: 7g*10 board/box, produced by Beijing Yucheng Health Technology Co., Ltd.
  Ilaprazole: 5mg*6 capsules/box, produced by Livzon Pharmaceutical Group Inc. Amoxicillin: 250mg*50 capsules/box, produced by Hainan General Sanyo Pharmaceutical Co., Ltd.
  Clarithromycin: 500mg*6 capsules/box, produced by Henan Fusen Pharmaceutical Co., Ltd.
  Furazolidone: 0.1g*28 pieces/bag, produced by Tianjin Lisheng Pharmaceutical Co., Ltd.
  Doxycycline: 0.1g*10 capsules/box, produced by Jiangsu Yongxin Pharmaceutical Co., Ltd.
  bismuth :55mg*36 capsules/box, produced by Shanxi Xinbaoyuan Pharmaceutical Co.,Ltd
  Arms: study group
Drug: IIaprazole, Amoxicillin/Clarithromycin/Furazolidone, Doxycycline, Bismuth — Ilaprazole: 5mg*6 capsules/box, produced by Livzon Pharmaceutical Group Inc. Amoxicillin: 250mg*50 capsules/box, produced by Hainan General Sanyo Pharmaceutical Co., Ltd.
  Clarithromycin: 500mg*6 capsules/box, produced by Henan Fusen Pharmaceutical Co., Ltd.
  Furazolidone: 0.1g*28 pieces/bag, produced by Tianjin Lisheng Pharmaceutical Co., Ltd.
  Doxycycline: 0.1g*10 capsules/box, produced by Jiangsu Yongxin Pharmaceutical Co., Ltd.
  bismuth :55mg*36 capsules/box, produced by Shanxi Xinbaoyuan Pharmaceutical Co.,Ltd
  Arms: control group
Drug: Yolk antibody and IIaprazole, Amoxicillin/ Clarithromycin/Furazolidone, Doxycycline — Yolk antibody: 7g*10 board/box, produced by Beijing Yucheng Health Technology Co., Ltd.
  Ilaprazole: 5mg*6 capsules/box, produced by Livzon Pharmaceutical Group Inc. Amoxicillin: 250mg*50 capsules/box, produced by Hainan General Sanyo Pharmaceutical Co., Ltd.
  Clarithromycin: 500mg*6 capsules/box, produced by Henan Fusen Pharmaceutical Co., Ltd.
  Furazolidone: 0.1g*28 pieces/bag, produced by Tianjin Lisheng Pharmaceutical Co., Ltd.
  Doxycycline: 0.1g*10 capsules/box, produced by Jiangsu Yongxin Pharmaceutical Co., Ltd.
  Arms: the case group
Drug: IIaprazole, Amoxicillin/ Clarithromycin/Furazolidone, Doxycycline, Bismuth — Ilaprazole: 5mg*6 capsules/box, produced by Livzon Pharmaceutical Group Inc. Amoxicillin: 250mg*50 capsules/box, produced by Hainan General Sanyo Pharmaceutical Co., Ltd.
  Clarithromycin: 500mg*6 capsules/box, produced by Henan Fusen Pharmaceutical Co., Ltd.
  Furazolidone: 0.1g*28 pieces/bag, produced by Tianjin Lisheng Pharmaceutical Co., Ltd.
  Doxycycline: 0.1g*10 capsules/box, produced by Jiangsu Yongxin Pharmaceutical Co., Ltd.
  bismuth :55mg*36 capsules/box, produced by Shanxi Xinbaoyuan Pharmaceutical Co.,Ltd
  Arms: the control group

SUMMARY:
Helicobacter pylori is an important pathogenic factor for gastrointestinal diseases such as gastritis, peptic ulcer, gastric mucosa-associated lymphoid tissue lymphoma and gastric cancer.However, with the increasing use of antibiotics, antibiotic resistance of Helicobacter pylori continues to rise. In this study, we used egg yolk antibody combined with bismuth quadruple therapy to treat patients with Helicobacter pylori infection, and observed the eradication rate of Helicobacter pylori, the relief of clinical symptoms and the incidence of adverse reactions.

DETAILED DESCRIPTION:
Background: Helicobacter pylori is an important pathogenic factor for gastrointestinal diseases such as gastritis, peptic ulcer, gastric mucosa-associated lymphoid tissue lymphoma and gastric cancer.However, with the increasing use of antibiotics, antibiotic resistance of Helicobacter pylori continues to rise. Therefore, it is of great significance to explore new methodsfor the treatment of Helicobacter pylori.

Methods: A total of 200 patients who failed to eradicate Helicobacter pylori were included and randomly divided into control group and study group. The research group was treated with egg yolk antibody combined with bismuth quadruple therapy, and the research group was treated with bismuth quadruple therapy for a total of 14 days. The eradication rate of Helicobacter pylori was calculated according to intention-to-treat and by-protocol analysis, and the symptom remission rate and adverse reactions were recorded during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years old, male or female;
2. Patients diagnosed with Hp infection;
3. Failure of Hp eradication therapy;
4. Although taking acid-suppressing drugs (PPI), the drug has been stopped for more than 2 weeks;
5. Those who have not used antibiotics and (or) bismuth in the past 4 weeks;
6. Understand and be willing to participate in this clinical trial and provide signed informed consent.

Exclusion Criteria:

1. Those with a history of allergy to drugs and egg yolk antibody products;
2. Those with severe heart, liver, lung and kidney insufficiency;
3. Those with a recent history of gastrointestinal bleeding, obstruction, perforation, tumor, and other serious organic diseases of the gastrointestinal tract;
4. Those with mental illness or mental disorder that cannot be expressed normally;
5. During the research period, those who are pregnant, breastfeeding, or have a childbearing plan recently;
6. There are other persons who are not suitable for clinical trials of drugs
7. No collaborators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | At four weeks after the completion of treatment (day 42±3)
  Detected by 13C-urea breath test (13C-UBT) or 14C-urea breath test (14-UBT), Eradication rate=(Number of successful eradication / total number of eradication)*100%

SECONDARY OUTCOMES:
Relief of clinical symptoms (Symptom relief rate) | After drug treatment (day 14±3) and during follow-up (day 42±3)
  Assessment by questionnaire: Symptom relief rate = (number of people with relief of symptoms/total number of people) *100%
Adverse events | After drug treatment (day 14±3)
  follow up to get the percentage of people with adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: SHA CHENG, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No